CLINICAL TRIAL: NCT03146416
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Evinacumab in Healthy Japanese and Caucasian Subjects
Brief Title: Study of Evinacumab (REGN1500) in Caucasian and in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: R1500-CL-1642
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evinacumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cohort 1 (Experimental): Evinacumab SC or placebo SC
  Interventions: Drug: Evinacumab; Drug: Placebo
- Cohort 2 (Experimental): Low dose regimen: evinacumab IV or placebo IV
  Interventions: Drug: Evinacumab; Drug: Placebo
- Cohort 3 (Experimental): High dose regimen: evinacumab IV or placebo IV
  Interventions: Drug: Evinacumab; Drug: Placebo
- Cohort 4 (Experimental): Evinacumab or placebo SC every week (QW) x 8 doses
  Interventions: Drug: Evinacumab; Drug: Placebo
- Cohort 5 (Experimental): Evinacumab or placebo SC x 1 dose
  Interventions: Drug: Evinacumab; Drug: Placebo

INTERVENTIONS:
Drug: Evinacumab — SC or IV administration of Evinacumab
  Other Names: REGN1500
Drug: Placebo — Matching placebo

SUMMARY:
The primary objective of the study is to compare the safety and tolerability of subcutaneous (SC) and intravenous (IV) doses of evinacumab in healthy Japanese and Caucasian subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or female Japanese and Caucasian volunteers ≥18 and ≤55 years of age at the screening visit.
* Japanese subjects must:

  1. Be first generation Japanese, defined as born in Japan and both biologic parents are ethnic Japanese
  2. Have maintained a Japanese lifestyle that has not significantly changed since leaving Japan, including having access to Japanese food and adhering to a Japanese diet.
* Caucasian subjects must be Caucasian of European or Latin American descent
* Modest elevations in LDL-C (≥100 mg/dL, but <160 mg/dL)

Key Exclusion Criteria:

* Significant concomitant illness
* Known allergy or sensitivity to monoclonal antibodies (mAbs)
* Previous exposure to anti-ANGPTL3 antibody
* Body mass index (BMI) >35 kg/m2 at the screening visit

Note: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Baseline up to week 31
Severity of TEAEs | Baseline up to week 31

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of evinacumab for geometric means of maximum (or peak) serum concentration (Cmax) | Up to Week 31
PK parameters of evinacumab for geometric means of Area under the curve (AUC) computed from time zero to the last measurable concentration (AUClast) | Up to Week 31
  single dose cohort
PK parameters of evinacumab for geometric means of AUC computed from time zero to the end of a dosing interval (AUCtau) | Up to Week 31
  following the first dose for the multiple dose cohorts
Ratio of Japanese versus Caucasian populations for geometric means of Cmax | Up to Week 31
Ratio of Japanese versus Caucasian populations for geometric means of AUClast | Up to Week 31
  single dose cohort
Ratio of Japanese versus Caucasian populations for geometric means of AUCtau | Up to Week 31
  following the first dose for the multiple dose cohorts
Absolute change from baseline over time in the Pharmacodynamic (PD) variable: Low-density lipoprotein cholesterol (LDL-C) | Up to Week 31
Absolute change from baseline over time in the PD variable: Total cholesterol | Up to Week 31
Absolute change from baseline over time in the PD variable: High-density lipoprotein cholesterol (HDL-C) | Up to Week 31
Absolute change from baseline over time in the PD variable: Triglycerides | Up to Week 31
Absolute change from baseline over time in the PD variable: non-HDL-C | Up to Week 31
Absolute change from baseline over time in the PD variable: lipoprotein a [Lp(a)] | Up to Week 31
Absolute change from baseline over time in the PD variable: apolipoprotein B [ApoB] | Up to Week 31
Absolute change from baseline over time in the PD variable: apolipoprotein A1 [ApoA1] | Up to Week 31
Absolute change from baseline over time in the PD variable: apolipoprotein C3 [ApoC3] | Up to Week 31
Absolute change from baseline over time in the PD variable: high-sensitivity C-reactive protein [hs-CRP] | Up to Week 31
Absolute change from baseline over time in the PD variable: Total Angiopoietin-like 3 (ANGPTL3) | Up to Week 31
Percent change from baseline over time in the PD variable: LDL-C | Up to Week 31
Percent change from baseline over time in the PD variable: Total cholesterol | Up to Week 31
Percent change from baseline over time in the PD variable: HDL-C | Up to Week 31
Percent change from baseline over time in the PD variable: Triglycerides | Up to Week 31
Percent change from baseline over time in the PD variable: non-HDL-C | Up to Week 31
Percent change from baseline over time in the PD variable: lipoprotein a [Lp(a)] | Up to Week 31
Percent change from baseline over time in the PD variable: apolipoprotein B [ApoB] | Up to Week 31
Percent change from baseline over time in the PD variable: apolipoprotein A1 [ApoA1] | Up to Week 31
Percent change from baseline over time in the PD variable: apolipoprotein C3 [ApoC3] | Up to Week 31
Percent change from baseline over time in the PD variable: high-sensitivity C-reactive protein [hs-CRP] | Up to Week 31
Percent change from baseline over time in the PD variable: Total (ANGPTL3) | Up to Week 31
Presence and titer of anti-evinacumab antibodies | Up to Week 31

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

REFERENCES:
- [Derived] Harada-Shiba M, Ali S, Gipe DA, Gasparino E, Son V, Zhang Y, Pordy R, Catapano AL. A randomized study investigating the safety, tolerability, and pharmacokinetics of evinacumab, an ANGPTL3 inhibitor, in healthy Japanese and Caucasian subjects. Atherosclerosis. 2020 Dec;314:33-40. doi: 10.1016/j.atherosclerosis.2020.10.013. Epub 2020 Oct 10. PMID 33130482